CLINICAL TRIAL: NCT03014453
Title: Gastroesophageal Reflux Poses a Potential Risk for Late Complications of BPD: A Prospective Study
Brief Title: GER Poses a Potential Risk for Late Complications of BPD
Status: Completed | Type: Observational
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Shucheng Zhang, Professor, Shengjing Hospital
Other Study IDs: A333-1
Record Dates: First submitted 2017-01-05; First posted 2017-01-09 (Estimated); Results first posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Gastroesophageal Reflux; Bronchopulmonary Dysplasia
MeSH Terms: conditions — Gastroesophageal Reflux; Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Bronchopulmonary dysplasia (BPD) is a common condition in the low birth weight infants. Although most of the BPD symptoms improved after a regular treatment in infancy, there are still a few late complications left such as the frequent respiratory symptoms, a slower weight gain and even sudden death. These late complications have made so much trouble to the healthcare of BPD infants. How to find the risk factors and to reduce the prevalence of these late symptoms becomes necessary. In this study, a cohort of BPD infants was observed with the late complications obtained by a monthly followed up for 18 months after discharge, the prevalence and risk factors of the late complications of BPD were analyzed by logistic regression. As one of the risk factors, GER was verified whether to play a critical role in these late complications.

ELIGIBILITY:
Inclusion Criteria:

* the extremely premature infants with bronchopulmonary dysplasia

Exclusion Criteria:

* other congenital malformations such as gastrointestinal and or neurogenic disease

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Extremely Premature Infants with Bronchopulmonary Dysplasia
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital, Shenyang, Liaoning, China

REFERENCES:
- [Background] Kalikkot Thekkeveedu R, Guaman MC, Shivanna B. Bronchopulmonary dysplasia: A review of pathogenesis and pathophysiology. Respir Med. 2017 Nov;132:170-177. doi: 10.1016/j.rmed.2017.10.014. Epub 2017 Oct 24. PMID 29229093
- [Background] Bonadies L, Zaramella P, Porzionato A, Muraca M, Baraldi E. Bronchopulmonary dysplasia: what's new on the horizon? Lancet Child Adolesc Health. 2018 Aug;2(8):549-551. doi: 10.1016/S2352-4642(18)30181-0. Epub 2018 Jun 27. No abstract available. PMID 30119711
- [Background] Papagianis PC, Pillow JJ, Moss TJ. Bronchopulmonary dysplasia: Pathophysiology and potential anti-inflammatory therapies. Paediatr Respir Rev. 2019 Apr;30:34-41. doi: 10.1016/j.prrv.2018.07.007. Epub 2018 Jul 29. PMID 30201135
- [Background] Perez Tarazona S, Solano Galan P, Bartoll Alguacil E, Alfonso Diego J. Bronchopulmonary dysplasia as a risk factor for asthma in school children and adolescents: A systematic review. Allergol Immunopathol (Madr). 2018 Jan-Feb;46(1):87-98. doi: 10.1016/j.aller.2017.02.004. Epub 2017 Jun 28. PMID 28668285
- [Background] Clyman RI. Patent ductus arteriosus, its treatments, and the risks of pulmonary morbidity. Semin Perinatol. 2018 Jun;42(4):235-242. doi: 10.1053/j.semperi.2018.05.006. Epub 2018 May 10. PMID 29958703
- [Background] Nagiub M, Kanaan U, Simon D, Guglani L. Risk Factors for Development of Pulmonary Hypertension in Infants with Bronchopulmonary Dysplasia: Systematic Review and Meta-Analysis. Paediatr Respir Rev. 2017 Jun;23:27-32. doi: 10.1016/j.prrv.2016.11.003. Epub 2016 Nov 22. PMID 28188008
- [Background] Vandenplas Y, Goyvaerts H, Helven R, Sacre L. Gastroesophageal reflux, as measured by 24-hour pH monitoring, in 509 healthy infants screened for risk of sudden infant death syndrome. Pediatrics. 1991 Oct;88(4):834-40. PMID 1896295
- [Background] Hassall E. Decisions in diagnosing and managing chronic gastroesophageal reflux disease in children. J Pediatr. 2005 Mar;146(3 Suppl):S3-12. doi: 10.1016/j.jpeds.2004.11.034. PMID 15758900
- [Background] Rosen R, Vandenplas Y, Singendonk M, Cabana M, DiLorenzo C, Gottrand F, Gupta S, Langendam M, Staiano A, Thapar N, Tipnis N, Tabbers M. Pediatric Gastroesophageal Reflux Clinical Practice Guidelines: Joint Recommendations of the North American Society for Pediatric Gastroenterology, Hepatology, and Nutrition and the European Society for Pediatric Gastroenterology, Hepatology, and Nutrition. J Pediatr Gastroenterol Nutr. 2018 Mar;66(3):516-554. doi: 10.1097/MPG.0000000000001889. PMID 29470322
- [Background] Cohen S, Bueno de Mesquita M, Mimouni FB. Adverse effects reported in the use of gastroesophageal reflux disease treatments in children: a 10 years literature review. Br J Clin Pharmacol. 2015 Aug;80(2):200-8. doi: 10.1111/bcp.12619. Epub 2015 Jun 11. PMID 25752807
- [Background] Shakir AK, Altaf MA. Azithromycin Induces Migrating Motor Complexes in Pediatric Patients Undergoing Antroduodenal Motility Studies. J Pediatr Pharmacol Ther. 2018 Sep-Oct;23(5):390-394. doi: 10.5863/1551-6776-23.5.390. PMID 30429693
- [Background] Stoll BJ, Hansen NI, Bell EF, Shankaran S, Laptook AR, Walsh MC, Hale EC, Newman NS, Schibler K, Carlo WA, Kennedy KA, Poindexter BB, Finer NN, Ehrenkranz RA, Duara S, Sanchez PJ, O'Shea TM, Goldberg RN, Van Meurs KP, Faix RG, Phelps DL, Frantz ID 3rd, Watterberg KL, Saha S, Das A, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Neonatal outcomes of extremely preterm infants from the NICHD Neonatal Research Network. Pediatrics. 2010 Sep;126(3):443-56. doi: 10.1542/peds.2009-2959. Epub 2010 Aug 23. PMID 20732945
- [Background] Parad RB, Davis JM, Lo J, Thomas M, Marlow N, Calvert S, Peacock JL, Greenough A. Prediction of respiratory outcome in extremely low gestational age infants. Neonatology. 2015;107(4):241-8. doi: 10.1159/000369878. Epub 2015 Mar 3. PMID 25765705
- [Derived] Wang LJ, Hu Y, Wang W, Zhang CY, Bai YZ, Zhang SC. Gastroesophageal Reflux Poses a Potential Risk for Late Complications of Bronchopulmonary Dysplasia: A Prospective Cohort Study. Chest. 2020 Oct;158(4):1596-1605. doi: 10.1016/j.chest.2020.05.523. Epub 2020 May 22. PMID 32450238

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The cohort study was conducted with BPD infants born≤32 weeks gestational age (GA) between January 2017 and July 2018 at Shengjing Hospital of China Medical University.The BPD was diagnosed at 36 weeks postmenstrual age (PMA) on the National Heart, Lung and Blood Institute classification and categorized as "mild, moderate or severe".
Groups:
- Extremely Premature Infants With Bronchopulmonary Dysplasia: Single arm-extremely premature infants with bronchopulmonary dysplasia
Period: Overall Study
Arm/Group | Extremely Premature Infants With Bronchopulmonary Dysplasia
Started | 187
Completed | 116
Not Completed | 71
Not completed — Lost to Follow-up | 12
Not completed — Discontinued GER | 3
Not completed — Excluded | 19
Not completed — Refused to take part in | 37

BASELINE CHARACTERISTICS:
Groups:
- Extremely Premature Infants With Bronchopulmonary Dysplasia: This observational cohort study was conducted with BPD infants born≤32 weeks gestational age (GA) at Shengjing Hospital of China Medical University neonatal intensive care unit (NICU). None of them received antacid medications, inhaled medications, or diuretics.
Arm/Group | Extremely Premature Infants With Bronchopulmonary Dysplasia
Number analyzed (Participants) | 116
Age, Customized [Number; unit: participants] — Gestational age at birth is reported
  participants
    gestational age>=30 week | 65
    gestational age<30 week | 51
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 72
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
birth weight [Count of Participants; unit: Participants]
  >1500g | 45
  <1500g | 71
1min Apgar [Count of Participants; unit: Participants] — 1 min Apgar score was described. If the 1min Apgar score <7, it was considered neonatal asphyxia，otherwise it was regarded as normal infant.
  Participants
    1min Apgar<7 | 27
    1 min Apgar>=7 | 89
Invasive ventilation [Count of Participants; unit: Participants] — Describes the duration of the use of invasive ventilation during hospitalization
  Participants
    Invasive ventilation>=7 days | 28
    Invasive ventilation<7 days | 88
Application of pulmonary surfactant [Count of Participants; unit: Participants] — Describes whether pulmonary surfactant has been used
  Participants
    yes | 76
    no | 40
Application of caffeine [Count of Participants; unit: Participants] — Describes whether caffeine therapy has been used
  Participants
    yes | 79
    no | 37
Ventilator-associated Pneumonia [Count of Participants; unit: Participants] — Cases of ventilator-associated pneumonia during hospitalization
  Participants
    yes | 55
    no | 61
patent ductus arteriosus [Count of Participants; unit: Participants] — Cases of patent ductus arteriosus
  Participants
    yes | 29
    no | 87
Gastroesophageal reflux [Count of Participants; unit: Participants] — The cases were diagnosed as gastroesophageal reflux by pH-MII and determination of gastric sodium ions．
  Participants
    No | 67
    Acid GER | 21
    DGER | 28

OUTCOME MEASURES:

1. Primary Outcome: the Late Complications of BPD Infants
Description: In all patients, complications were evaluated via questionnaires at 3, 6, 9 and 12 months corrected for premature age, including respiratory symptoms (including home respiratory support, respiratory medication administration, cough without cold at least once per week, re-hospitalization due to respiratory diseases), vomiting when feeding, hypoxic ischemic injury, retinopathy of prematurity, rehospitalization and sudden death.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Extremely Premature Infants With Bronchopulmonary Dysplasia
Number analyzed (Participants) | 116
Participants
  respiratory symptoms | 57
  Vomiting when feeding | 45
  retinopathy of prematurity | 30
  hypoxic ischemic injury | 4
  sudden infant death syndrome | 1
  rehospitalization | 31

ADVERSE EVENTS:
Time Frame: 18 month
Arm/Group | Extremely Premature Infants With Bronchopulmonary Dysplasia
All-Cause Mortality (participants affected / at risk) | 1/116
Serious Adverse Events (participants affected / at risk) | 64/116
Other Adverse Events (participants affected / at risk) | 69/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extremely Premature Infants With Bronchopulmonary Dysplasia (N=116)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 10 (116)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (116)
cyanosis (Respiratory, thoracic and mediastinal disorders) | 10 (116)
intermittent apnea (Respiratory, thoracic and mediastinal disorders) | 5 (116)
retinopathy of prematurity (Eye disorders) | 30 (116)
hypoxic ischemic injury (Nervous system disorders) | 4 (116)
Re-hospitalization (Respiratory, thoracic and mediastinal disorders) | 31 (116)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extremely Premature Infants With Bronchopulmonary Dysplasia (N=116)
cough without cold (Respiratory, thoracic and mediastinal disorders) | 44 (116) — cough without cold at least once per week
Vomiting when feeding (General disorders) | 45 (116)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-24): https://cdn.clinicaltrials.gov/large-docs/53/NCT03014453/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-24): https://cdn.clinicaltrials.gov/large-docs/53/NCT03014453/ICF_001.pdf